CLINICAL TRIAL: NCT03096704
Title: Vitamine D Deficiency in Slow Transit Time Constipation
Brief Title: Vitamine d Dosage and Constipation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, alba panarese, principal investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 29
Record Dates: First submitted 2017-03-26; First posted 2017-03-30 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Vitamine d Dosage in Slow Transit Time Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- slow transit time constipation
  Interventions: Diagnostic Test: vitamine d dosage

INTERVENTIONS:
Diagnostic Test: vitamine d dosage — dosage of vitamine D in slow transit time constipation

SUMMARY:
Vitamine d dosage in important to define nutritional status and bone metabolism. For patients with intestinal disorders it is important to establish the intestinal absorptive function.

It is important to establish the absorption of vitamin D which correlate with different biological activity and bone metabolism, immune function and the communication between the cells.

DETAILED DESCRIPTION:
Constipation is a disease that involves poor intestinal functioning. The reduced intestinal motility slows down intestinal function. Up to make lower the dosage of vitamin D. Vitamin D helps many cellular activities and enhances the action of tissue,Its Your dosage allows you to evaluate the efficacy of intestinal function and to better understand its severity.

ELIGIBILITY:
Inclusion Criteria:

* slow transit time constipation

Exclusion Criteria:

* drugs assumption comorbidity

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: observational prospective study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-04-30 (Estimated); Study Completion 2017-05-15 (Estimated)

PRIMARY OUTCOMES:
dosage of vitamine D | 4 months
  dosage of vitamine d in slow transit time constipation

CONTACTS AND LOCATIONS:
Locations (1):
- Alba Panarese, Noci, Apulia, Italy

IPD SHARING:
Plan to Share IPD: Undecided